CLINICAL TRIAL: NCT05257226
Title: Both Short- and Long-term Outcome Differences According to Patient Frailty
Status: Recruiting | Type: Observational
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Department of Gastroenterological Surgery, Kochi University
Other Study IDs: Bos study
Record Dates: First submitted 2022-02-01; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: frailty — questionaire

SUMMARY:
The evaluation for cancer treatment successful has been used by overall survival rate and/or postoperative complications, especially surgical area. Now postoperative QOL has been more importantly required. Therefore this study was conduced to investigate the association between postoperative outcomes and patients frailty.

ELIGIBILITY:
Inclusion Criteria:

* surgical patients

Exclusion Criteria:

* a body weight loss of >10% during the 6 months before surgery; the presence of distant metastases; or seriously impaired function of vital organs because of respiratory, renal, or heart disease

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: surgically treated patients for gastroenterological diseases
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative short-term outcomes | up to 24 weeks
  postoperative complications

SECONDARY OUTCOMES:
postoperative long-term outcomes | 5 year
  survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Takehiro Okabayashi, Kochi, Japan

IPD SHARING:
Plan to Share IPD: No